CLINICAL TRIAL: NCT04469465
Title: A Phase 3 Study of Danicopan (ALXN2040) as Add-on Therapy to a C5 Inhibitor (Eculizumab or Ravulizumab) in Patients With Paroxysmal Nocturnal Hemoglobinuria Who Have Clinically Evident Extravascular Hemolysis (EVH)
Brief Title: Danicopan as Add-on Therapy to a C5 Inhibitor in Paroxysmal Nocturnal Hemoglobinuria (PNH) Participants Who Have Clinically Evident Extravascular Hemolysis (EVH)(ALPHA)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ALXN2040-PNH-301; 2019-003829-18 (EudraCT Number)
Record Dates: First submitted 2020-07-09; First posted 2020-07-14 (Actual); Results first posted 2023-07-24 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-04

CONDITIONS: Paroxysmal Nocturnal Hemoglobinuria
Keywords: Paroxysmal Nocturnal Hemoglobinuria (PNH); Extravascular Hemolysis (EVH); Factor D inhibitor; Complement; Danicopan; C5 inhibitor
MeSH Terms: conditions — Hemoglobinuria, Paroxysmal; Hemolysis | interventions — danicopan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Danicopan + C5 Inhibitor (Experimental): Participants will receive danicopan, in addition to their C5 inhibitor therapy, for 24 weeks (12 weeks in Treatment Period 1, followed by 12 weeks in Treatment Period 2).
  Interventions: Drug: Danicopan; Drug: C5 Inhibitor
- Placebo + C5 Inhibitor (Placebo Comparator): Participants will receive placebo, in addition to their C5 inhibitor therapy, for 12 weeks during Treatment Period 1. At Week 12, participants randomized to receive placebo will be switched to danicopan for an additional 12 weeks (Treatment Period 2).
  Interventions: Drug: Placebo; Drug: C5 Inhibitor

INTERVENTIONS:
Drug: Danicopan — Oral tablet
  Other Names: ALXN2040
  Arms: Danicopan + C5 Inhibitor
Drug: Placebo — Oral tablet
  Arms: Placebo + C5 Inhibitor
Drug: C5 Inhibitor — Participants will continue to receive their ongoing C5 inhibitor (eculizumab or ravulizumab) therapy according to their usual dose and schedule.

SUMMARY:
The main objective of this study is to evaluate the efficacy of danicopan as add-on therapy to a complement component 5 (C5) inhibitor (eculizumab or ravulizumab) in participants with PNH who have clinically evident EVH.

DETAILED DESCRIPTION:
This is a multiple-region, randomized, double-blind, placebo controlled, multiple-dose, study in participants with PNH who have clinically evident EVH on a C5 inhibitor (eculizumab or ravulizumab).

Participants will be randomized to receive danicopan or placebo, in a 2:1 ratio for 12 weeks (Treatment Period 1) in addition to their C5 inhibitor (eculizumab or ravulizumab) therapy. At Week 12, participants randomized to receive placebo will be switched to danicopan in addition to their C5 inhibitor for an additional 12 weeks (Treatment Period 2) and participants randomized to danicopan will continue on danicopan for an additional 12 weeks, while remaining on their ongoing C5 inhibitor therapy.

At the end of the 2 treatment periods (Week 24), participants may enter a Long-Term Extension (LTE) Period and continue to receive danicopan in addition to their C5 inhibitor therapy. The Long-Term Extension period will consist of a first year of LTE(Year1) and a second year of optional LTE(Year2).All patients will complete 72 weeks of LTE(Year 1) assessments. After Week 72 (at the end of the first year of LTE), patients have the choice to complete participation in this study or continue to the optional second year (Year2) of LTE.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of PNH
* Clinically Evident EVH defined by:

  * Anemia (Hgb ≤9.5 gram/deciliter) with absolute reticulocyte count ≥120 x 10^9/liter
* Receiving an approved C5 inhibitor for at least 6 months prior to Day 1
* Platelet count ≥30,000/microliters (µL)
* Absolute neutrophil counts ≥500/μL
* Documentation of/or willingness to receive vaccinations for N. meningiditis and prophylactic antibiotics as required

Exclusion Criteria:

* History of a major organ transplant or hematopoietic stem cell transplantation (HSCT)
* Participants with known aplastic anemia or other bone marrow failure that requires HSCT or other therapies including anti-thymocyte globulin and/or immunosuppressants
* Known or suspected complement deficiency
* Laboratory abnormalities at screening, including:

  * Alanine aminotransferase >2 x ULN (>3 x ULN in case of patients with documented liver iron overload defined by serum ferratin values

    * 500 ng/ML)
  * Direct bilirubin >2 x ULN (unless due to EVH or documented Gilbert's Syndrome)
* Current evidence of biliary cholestasis
* Estimated glomerular filtration rate of <30 milliliters/minute/1.73 meter squared and/or are on dialysis
* Evidence of human immunodeficiency virus, hepatitis B, or active hepatitis C infection at screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2020-12-16 (Actual); Primary Completion 2022-06-29 (Actual); Study Completion 2024-01-16 (Actual)

CONTACTS AND LOCATIONS:
Locations (59):
- United States (7):
  - Research Site, Los Angeles, California
  - Research Site, Weston, Florida
  - Research Site, Chicago, Illinois
  - Research Site, Kalamazoo, Michigan
  - Research Site, New York, New York
  - Research Site, Dallas, Texas
  - Research Site, Milwaukee, Wisconsin
- Brazil (5):
  - Research Site, Belém
  - Research Site, Curitiba
  - Research Site, Goiânia
  - Research Site, Porto Alegre
  - Research Site, Rio de de Janeiro
- Research Site, Toronto, Ontario, Canada
- Research Site, Brno, Czechia
- France (4):
  - Research Site, Lille
  - Research Site, Paris
  - Research Site, Pessac
  - Research Site, Pierre-Bénite
- Research Site, Ulm, Germany
- Greece (2):
  - Research Site, Athens
  - Research Site, Thessaloniki
- Israel (2):
  - Research Site, Haifa
  - Research Site, Jerusalem
- Italy (6):
  - Research Site, Avellino
  - Research Site, Bassano del Grappa
  - Research Site, Florence
  - Research Site, Milan
  - Research Site, Reggio Calabria
  - Research Site, Roma
- Japan (12):
  - Research Site, Bunkyō City
  - Research Site, Fukuoka
  - Research Site, Kashiwa-shi
  - Research Site, Kyoto
  - Research Site, Nagakute-shi
  - Research Site, Ogaki-shi
  - Research Site, Osaka
  - Research Site, Sayama
  - Research Site, Shibuya-ku
  - Research Site, Tanabe-shi
  - Research Site, Toyoake-shi
  - Research Site, Tsukuba
- Malaysia (3):
  - Research Site, Kota Kinabalu
  - Research Site, Kuching
  - Research Site, Miri
- Research Site, Maastricht, Netherlands
- Research Site, Gdansk, Poland
- South Korea (3):
  - Research Site, Daejeon
  - Research Site, Seoul
  - Research Site, Suwon
- Spain (5):
  - Research Site, Barcelona
  - Research Site, Las Palmas de Gran Canaria
  - Research Site, Madrid
  - Research Site, Majadahonda
  - Research Site, Seville
- Research Site, Taipei, Taiwan
- Research Site, Bangkok, Thailand
- United Kingdom (3):
  - Research Site, Airdrie
  - Research Site, Leeds
  - Research Site, London

REFERENCES:
- [Result] Lee JW, Griffin M, Kim JS, Lee Lee LW, Piatek C, Nishimura JI, Carrillo Infante C, Jain D, Liu P, Filippov G, Sicre de Fontbrune F, Risitano A, Kulasekararaj AG; ALXN2040-PNH-301 Investigators. Addition of danicopan to ravulizumab or eculizumab in patients with paroxysmal nocturnal haemoglobinuria and clinically significant extravascular haemolysis (ALPHA): a double-blind, randomised, phase 3 trial. Lancet Haematol. 2023 Dec;10(12):e955-e965. doi: 10.1016/S2352-3026(23)00315-0. PMID 38030318
- [Derived] Kulasekararaj A, Griffin M, Piatek C, Shammo J, Nishimura JI, Patriquin C, Schrezenmeier H, Barcellini W, Panse J, Gaya A, Patel Y, Liu P, Filippov G, Sicre de Fontbrune F, Risitano A, Lee JW. Long-term efficacy and safety of danicopan as add-on therapy to ravulizumab or eculizumab in PNH with significant EVH. Blood. 2025 Feb 20;145(8):811-822. doi: 10.1182/blood.2024026299. PMID 39700502
- See also: Danicopan (ACH-4471) in Untreated Patients with Paroxysmal Nocturnal Hemoglobinuria (PNH) Phase 2, Open-label, Proof of Concept Study of the Oral, Small Molecule Factor D Inhibitor — https://library.ehaweb.org/eha/2019/24th/267447/peter.browett.a.phase.2.open
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=ALXN2040-PNH-301&attachmentIdentifier=5f3bdb66-e572-42a3-9aff-2abeca73c5f3&fileName=Synopsis_-_ALXN2040-PNH-301_Final_CSR_Redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study consists of 2 treatment periods and a long-term extension period.
Groups:
- Danicopan-Danicopan: Participants received danicopan TID for 12 weeks, in addition to their background ravulizumab or eculizumab therapy, during TP1. Participants continued to receive danicopan TID for an additional 12 weeks, in addition to their background ravulizumab or eculizumab therapy, during TP2. After completing TP2 (Week 24), participants entered the LTE for 2 years at the same danicopan dose received at Week 24, in addition to their background ravulizumab or eculizumab therapy.
- Placebo-Danicopan: Participants received placebo TID for 12 weeks, in addition to their background ravulizumab or eculizumab therapy, during TP1. At the end of Week 12, participants were switched to receive danicopan TID for 12 weeks, in addition to their background ravulizumab or eculizumab therapy, during TP2. After completing TP2 (Week 24), participants entered the LTE for 2 years at the same danicopan dose received at Week 24, in addition to their background ravulizumab or eculizumab therapy.
Period: Treatment Period 1 (TP1)
Arm/Group | Danicopan-Danicopan | Placebo-Danicopan
Started | 57 | 29
Received at Least 1 Dose of Study Drug (Full Analysis Set/Safety Set) | 57 | 29
Interim Efficacy Analysis Set (Per the prespecified plan for interim analysis, the first 75% of randomized participants formed the Interim Analysis Set for efficacy analysis.) | 42 | 21
Completed (Completed TP1) | 55 | 27
Not Completed | 2 | 2
Not completed — Adverse Event | 2 | 1
Not completed — Withdrawal by Subject | 0 | 1
Period: Treatment Period 2 (TP2)
Arm/Group | Danicopan-Danicopan | Placebo-Danicopan
Started | 55 | 27
Received at Least 1 Dose of Study Drug (Full Analysis Set/Safety Set) | 55 | 27
Completed | 54 | 26
Not Completed | 1 | 1
Not completed — Adverse Event | 1 | 1
Period: Long-Term Extension (LTE)
Arm/Group | Danicopan-Danicopan | Placebo-Danicopan
Started | 54 | 26
Received at Least 1 Dose of Study Drug (Safety Set) | 54 | 26
Completed | 46 | 24
Not Completed | 8 | 2
Not completed — Withdrawal by Subject | 3 | 0
Not completed — Physician Decision | 3 | 0
Not completed — Noncompliance with study intervention | 1 | 0
Not completed — Death | 0 | 1
Not completed — Adverse Event | 1 | 1

BASELINE CHARACTERISTICS:
Population: Full Analysis Set: all enrolled participants who were randomized to either the danicopan or placebo treatment group.
Groups:
- Danicopan-Danicopan: Participants received danicopan TID for 12 weeks, in addition to their background ravulizumab or eculizumab therapy, during TP1. Participants continued to receive danicopan TID for an additional 12 weeks, in addition to their background ravulizumab or eculizumab therapy, during TP2. After completing TP2 (Week 24), participants entered the long-term extension (LTE) for 2 years at the same danicopan dose received at Week 24, in addition to their background ravulizumab or eculizumab therapy.
- Total: Total of all reporting groups
Arm/Group | Danicopan-Danicopan | Placebo-Danicopan | Total
Number analyzed (Participants) | 57 | 29 | 86
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.8 (17.00) | 52.9 (14.34) | 52.8 (16.07)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 20 | 54
  Male | 23 | 9 | 32
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 1 | 7
  Not Hispanic or Latino | 46 | 24 | 70
  Unknown or Not Reported | 5 | 4 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 22 | 10 | 32
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 28 | 14 | 42
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 5 | 9
Hemoglobin (Hgb) [Mean (Standard Deviation); unit: g/L] — g/L = grams/liter
  g/L | 76.7 (9.47) | 78.9 (10.11) | 77.5 (9.69)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Hgb at Week 12
Description: Baseline was defined as the lowest Hgb value observed between and including Screening and Day 1. The least square (LS) mean and standard error (SE) were produced using mixed-effect model for repeated measures (MMRM). Hgb values collected within 4 weeks after transfusion were not included in the MMRM.
Time Frame: Baseline, Week 12
Population: Interim Efficacy Analysis Set: Per the prespecified plan for interim analysis, the first 75% of enrolled participants that were randomized to either the danicopan or placebo treatment group. Full Analysis Set: All enrolled participants that were randomized to either the danicopan or placebo treatment group. Here, 'Overall number of participants analyzed' = participants evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: g/L
Groups:
- Danicopan (TP1): Participants received danicopan TID for 12 weeks, in addition to their background ravulizumab or eculizumab therapy, during TP1.
- Placebo (TP1): Participants received placebo TID for 12 weeks, in addition to their background ravulizumab or eculizumab therapy, during TP1.
Arm/Group | Danicopan (TP1) | Placebo (TP1)
Number analyzed (Participants) | 57 | 28
g/L
  Interim Efficacy Analysis: number analyzed (Participants) | 42 | 21
  Interim Efficacy Analysis | 29.40 (2.107) | 4.96 (3.128)
  Full Analysis | 28.08 (1.957) | 4.62 (3.018)
Statistical Analysis 1: Comparison: Danicopan (TP1) vs Placebo (TP1); Interim Efficacy Analysis; Test type: Superiority; p = 0.0007, Re-randomization Test
Statistical Analysis 2: Comparison: Danicopan (TP1) vs Placebo (TP1); Full Analysis; Test type: Superiority; p = 0.0007, Re-randomization Test
Statistical Analysis 3: Comparison: Danicopan (TP1) vs Placebo (TP1); Interim Efficacy Analysis; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 24.44, 95% CI 2-sided [16.90 to 31.99], Standard Error of Mean 3.751
Statistical Analysis 4: Comparison: Danicopan (TP1) vs Placebo (TP1); Full Analysis; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Difference = 23.46, 95% CI 2-sided [16.31 to 30.61], Standard Error of Mean 3.585

2. Secondary Outcome: Percentage of Participants With Hgb Increase of ≥2 Grams/Deciliter (g/dL) (≥20 g/L) From Baseline in the Absence of Transfusion at Week 12
Description: The criterion was defined as ≥20 g/L increase in Hgb from Baseline to Week 12 and remaining transfusion free during the 12-Week TP1. Participants who withdrew from the study early during the 12-Week TP1 or had missing Hgb value at Week 12 were considered as not achieving the criterion.
Time Frame: Week 12
Population: Interim Efficacy Analysis Set: Per the prespecified plan for interim analysis, the first 75% of enrolled participants that were randomized to either the danicopan or placebo treatment group. Full Analysis Set: All enrolled participants that were randomized to either the danicopan or placebo treatment group.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Danicopan (TP1) | Placebo (TP1)
Number analyzed (Participants) | 57 | 29
percentage of participants
  Interim Efficacy Analysis: number analyzed (Participants) | 42 | 21
  Interim Efficacy Analysis | 59.5 [43.28 to 74.37] | 0 [0.00 to 16.11]
  Full Analysis | 54.4 [40.66 to 67.64] | 0 [0.00 to 11.94]

3. Secondary Outcome: Percentage of Participants With Transfusion Avoidance Through Week 12
Description: Participants achieved transfusion avoidance if they remained transfusion free and did not require a transfusion as per protocol-specified guidelines from Week 1 through Week 12. Participants who discontinued study treatment early before Week 12 were considered as not achieving transfusion avoidance.
Time Frame: Week 12
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Danicopan (TP1) | Placebo (TP1)
Number analyzed (Participants) | 57 | 29
percentage of participants
  Interim Efficacy Analysis: number analyzed (Participants) | 42 | 21
  Interim Efficacy Analysis | 83.3 [68.64 to 93.03] | 38.1 [18.11 to 61.56]
  Full Analysis | 78.9 [66.11 to 88.62] | 27.6 [12.73 to 47.24]

4. Secondary Outcome: Change From Baseline in Functional Assessment of Chronic Illness Therapy (FACIT) Fatigue Score at Week 12
Description: The FACIT-Fatigue was 13-item questionnaire scored on a 5-point Likert scale (0 = not at all, 4 = very much) that assesses self-reported fatigue and its impact on daily activities and function. Total scores range from 0 to 52 with higher score indicating less fatigue and better health-related quality of life. LS mean and SE were produced using MMRM.
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Danicopan (TP1) | Placebo (TP1)
Number analyzed (Participants) | 57 | 28
units on a scale
  Interim Efficacy Analysis: number analyzed (Participants) | 42 | 21
  Interim Efficacy Analysis | 7.97 (1.128) | 1.85 (1.581)
  Full Analysis: number analyzed (Participants) | 56 | 28
  Full Analysis | 8.13 (0.919) | 2.35 (1.289)

5. Secondary Outcome: Change From Baseline in Absolute Reticulocyte Count at Week 12
Description: LS mean and SE were produced using MMRM.
Time Frame: Baseline, Week 12
Population: Interim Efficacy Analysis Set: Per the prespecified plan for interim analysis, the first 75% of enrolled participants that were randomized to either the danicopan or placebo treatment group. Full Analysis Set: All enrolled participants that were randomized to either the danicopan or placebo treatment group. Here, 'Overall number of participants analyzed' and 'Number Analyzed' = participants evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: 10^12 cells/L
Arm/Group | Danicopan (TP1) | Placebo (TP1)
Number analyzed (Participants) | 57 | 26
10^12 cells/L
  Interim Efficacy Analysis: number analyzed (Participants) | 42 | 20
  Interim Efficacy Analysis | -0.0838 (0.00893) | 0.0035 (0.01268)
  Full Analysis | -0.0925 (0.00816) | -0.0008 (0.01184)

6. Secondary Outcome: Change in the Number of Red Blood Cell (RBC) Units Transfused From 24 Weeks Prior to Initiation of Treatment to Post 24 Weeks of Treatment
Time Frame: 24 weeks prior to initiation of treatment to 24 weeks post initiation of treatment
Population: Full Analysis Set: All enrolled participants that were randomized to the danicopan treatment group. Here, 'Overall Number of Participants Analyzed' signifies those participants who received danicopan who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: RBC units
Groups:
- Danicopan-Danicopan (TP2): Participants received danicopan TID for 12 weeks, in addition to their background ravulizumab or eculizumab therapy, during TP1. Participants continued to receive danicopan TID for an additional 12 weeks, in addition to their background ravulizumab or eculizumab therapy, during TP2.
Arm/Group | Danicopan-Danicopan (TP2)
Number analyzed (Participants) | 55
RBC units | -2.7 (4.86)

7. Secondary Outcome: Change in Number of Transfusion Instances From 24 Weeks Prior to Initiation of Treatment to Post 24 Weeks of Treatment
Time Frame: 24 weeks prior to initiation of treatment to 24 weeks post initiation of treatment
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: transfusion instances
Arm/Group | Danicopan-Danicopan (TP2)
Number analyzed (Participants) | 55
transfusion instances | -1.5 (2.41)

8. Secondary Outcome: Percentage of Participants With Transfusion Avoidance Through Week 24
Description: Participants achieved transfusion avoidance if they remained transfusion free and did not require a transfusion as per protocol-specified guidelines from Week 1 through Week 24. Participants who discontinued study treatment early before Week 24 were considered as not achieving transfusion avoidance.
Time Frame: 24 weeks
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Danicopan-Danicopan (TP2)
Number analyzed (Participants) | 55
percentage of participants | 69.1 [55.19 to 80.86]

9. Secondary Outcome: Change in the Number of RBC Units Transfused From 12 Weeks Prior to Initiation of Treatment to Post 12 Weeks of Treatment
Description: LS mean and SE were produced using analysis of covariance (ANCOVA).
Time Frame: 12 weeks prior to initiation of treatment to 12 weeks post initiation of treatment
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: RBC units
Arm/Group | Danicopan (TP1) | Placebo (TP1)
Number analyzed (Participants) | 57 | 29
RBC units
  Interim Efficacy Analysis: number analyzed (Participants) | 42 | 21
  Interim Efficacy Analysis | -1.48 (0.271) | -0.18 (0.383)
  Full Analysis | -1.44 (0.212) | -0.14 (0.297)

10. Secondary Outcome: Change in Number of Transfusion Instances From 12 Weeks Prior to Initiation of Treatment to Post 12 Weeks of Treatment
Description: LS mean and SE were produced using ANCOVA.
Time Frame: 12 weeks prior to initiation of treatment to post 12 weeks of treatment (24 weeks)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: transfusion instances
Arm/Group | Danicopan (TP1) | Placebo (TP1)
Number analyzed (Participants) | 57 | 29
transfusion instances
  Interim Efficacy Analysis: number analyzed (Participants) | 42 | 21
  Interim Efficacy Analysis | -0.92 (0.174) | -0.21 (0.246)
  Full Analysis | -0.91 (0.138) | -0.11 (0.193)

11. Secondary Outcome: Change From Baseline FACIT Fatigue Scores at Week 24
Description: as for outcome 4
Time Frame: Baseline, Week 24
Population: Full Analysis Set: All enrolled participants that were randomized to either the danicopan or placebo treatment group. Here, 'Overall Number of Participants Analyzed' signifies those participants who were evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- Danicopan-Danicopan: Participants received danicopan TID for 12 weeks, in addition to their background ravulizumab or eculizumab therapy, during TP1. Participants continued to receive danicopan TID for an additional 12 weeks, in addition to their background ravulizumab or eculizumab therapy, during TP2.
- Placebo-Danicopan: Participants received placebo TID for 12 weeks, in addition to their background ravulizumab or eculizumab therapy, during TP1. At the end of Week 12, participants were switched to receive danicopan TID for 12 weeks, in addition to their background ravulizumab or eculizumab therapy, during TP2.
Arm/Group | Danicopan-Danicopan | Placebo-Danicopan
Number analyzed (Participants) | 52 | 27
units on a scale | 6.21 (1.046) | 5.64 (1.921)

12. Secondary Outcome: Percentage of Participants With Hgb Stabilization During Last 12 Weeks of Treatment in Participants Receiving 24 Weeks of Danicopan
Description: The criterion was defined as Hgb stabilization avoidance of a >1 g/dL (>10 g/L) decrease in Hgb level at Week 24 from Week 12. Participants with transfusions within 4 weeks prior to Week 24 were considered as not meeting Hgb stabilization regardless of the actual value observed at Week 24.
Time Frame: Week 12 to Week 24
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Danicopan-Danicopan
Number analyzed (Participants) | 55
percentage of participants | 58.2 [44.11 to 71.35]

13. Secondary Outcome: Percentage of Participants With Hgb Increase of ≥2 g/dL (≥ 20 g/L) From Baseline in the Absence of Transfusion at Week 24
Description: The criterion was defined as ≥20 g/L increase in Hgb from Baseline to Week 24 and remaining transfusion free during the 12-Week TP2. Participants who withdrew from the study early during the 12-Week TP2 or had missing Hgb value at Week 24 were considered as not achieving the criterion.
Time Frame: Week 24
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Danicopan-Danicopan
Number analyzed (Participants) | 55
percentage of participants | 41.8 [28.65 to 55.89]

14. Secondary Outcome: Change From Baseline in Total and Direct Bilirubin at Week 12
Description: Baseline was defined as the last non-missing value prior to first dose of study intervention. LS mean and SE were produced using MMRM.
Time Frame: Baseline, Week 12
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: micromoles/L
Arm/Group | Danicopan (TP1) | Placebo (TP1)
Number analyzed (Participants) | 57 | 29
micromoles/L
  Total Bilirubin (Interim Efficacy Analysis): number analyzed (Participants) | 42 | 21
  Total Bilirubin (Interim Efficacy Analysis) | -9.77 (1.692) | -2.15 (2.377)
  Direct Bilirubin (Interim Efficacy Analysis): number analyzed (Participants) | 42 | 21
  Direct Bilirubin (Interim Efficacy Analysis) | -2.88 (0.357) | 0.30 (0.503)
  Total Bilirubin (Full Analysis) | -11.55 (1.541) | -1.42 (2.172)
  Direct Bilirubin (Full Analysis) | -2.85 (0.317) | 0.17 (0.447)

15. Secondary Outcome: Change From Baseline in Paroxysmal Nocturnal Hemoglobinuria (PNH) RBC Clone Size at Week 12
Description: The PNH clone size refers to the percentage of PNH-affected cells versus normal cells within the total cell population. Baseline was defined as the last non-missing value prior to first dose of study intervention. LS mean and SE were produced using MMRM.
Time Frame: Baseline, Week 12
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: percentage of the total cell population
Arm/Group | Danicopan (TP1) | Placebo (TP1)
Number analyzed (Participants) | 37 | 24
percentage of the total cell population
  Interim Efficacy Analysis: number analyzed (Participants) | 14 | 8
  Interim Efficacy Analysis | 24.60 (4.180) | -3.04 (5.864)
  Full Analysis | 26.35 (2.369) | -0.18 (2.960)

16. Secondary Outcome: Change From Baseline in Complement Component 3 Fragment Deposition (C3d PNH Type 3 Cells) on PNH RBCs at Week 12
Description: as for outcome 14
Time Frame: Baseline, Week 12
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: percentage of the total cell population
Arm/Group | Danicopan (TP1) | Placebo (TP1)
Number analyzed (Participants) | 56 | 26
percentage of the total cell population
  Interim Efficacy Analysis: number analyzed (Participants) | 23 | 10
  Interim Efficacy Analysis | -15.06 (2.824) | 0.89 (4.394)
  Full Analysis | -19.00 (1.814) | 0.68 (2.690)

17. Secondary Outcome: Change From Baseline in Lactate Dehydrogenase at Week 12
Description: Baseline was defined as the average of all available assessments prior to the first dose of study intervention. LS mean and SE were produced using MMRM.
Time Frame: Baseline, Week 12
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: units/L
Arm/Group | Danicopan (TP1) | Placebo (TP1)
Number analyzed (Participants) | 56 | 28
units/L
  Interim Efficacy Analysis: number analyzed (Participants) | 42 | 20
  Interim Efficacy Analysis | -23.49 (8.287) | -2.92 (11.914)
  Full Analysis | -25.60 (7.932) | -16.92 (11.380)

18. Secondary Outcome: Percentage of Participants With Hgb Normalization at Week 12
Description: Hgb normalization was defined as Hgb value above lower limit of normal (LLN) reference range. For male, the LLN was 125 g/L, for female, the LLN was 110 g/L. Participants with transfusions within 4 weeks prior to Week 12 were considered as not meeting Hgb normalization regardless of actual value observed at Week 12.
Time Frame: Week 12
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Danicopan (TP1) | Placebo (TP1)
Number analyzed (Participants) | 57 | 29
percentage of participants
  Interim Efficacy Analysis: number analyzed (Participants) | 42 | 21
  Interim Efficacy Analysis | 28.6 [15.72 to 44.58] | 0 [0.00 to 16.11]
  Full Analysis | 26.3 [15.54 to 39.66] | 0 [0.00 to 11.94]

19. Secondary Outcome: Percentage of Participants With Hgb Normalization at Week 24
Description: Hgb normalization was defined as Hgb value above LLN reference range. For male, the LLN was 125 g/L, for female, the LLN was 110 g/L. Participants with transfusions within 4 weeks prior to Week 24 were considered as not meeting Hgb normalization regardless of actual value observed at Week 24.
Time Frame: Week 24
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Danicopan-Danicopan
Number analyzed (Participants) | 55
percentage of participants | 20.0 [10.43 to 32.97]

ADVERSE EVENTS:
Time Frame: Baseline (Day 1) up to 30 days after last dose of study drug (approximately 2 years)
Description: The Safety Set included all participants that received at least 1 dose of study drug (danicopan or placebo).
Groups:
- Danicopan (TP1): Participants received danicopan TID for 12 weeks, in addition to their background ravulizumab or eculizumab therapy, during TP.
- Danicopan-Danicopan (TP2): Participants continued to receive danicopan TID for an additional 12 weeks, in addition to their background ravulizumab or eculizumab therapy, during TP2.
- Placebo-Danicopan (TP2): At the end of Week 12, participants were switched to receive danicopan TID for 12 weeks, in addition to their background ravulizumab or eculizumab therapy, during TP2.
- Danicopan-Danicopan (LTE); Placebo-Danicopan (LTE): After completing TP2 (Week 24), participants entered the LTE for 2 years at the same danicopan dose received at Week 24, in addition to their background ravulizumab or eculizumab therapy.
Arm/Group | Danicopan (TP1) | Placebo (TP1) | Danicopan-Danicopan (TP2) | Placebo-Danicopan (TP2) | Danicopan-Danicopan (LTE) | Placebo-Danicopan (LTE)
All-Cause Mortality (participants affected / at risk) | 0/57 | 0/29 | 0/55 | 0/27 | 0/54 | 1/26
Serious Adverse Events (participants affected / at risk) | 3/57 | 2/29 | 3/55 | 6/27 | 7/54 | 6/26
Other Adverse Events (participants affected / at risk) | 43/57 | 18/29 | 40/55 | 18/27 | 48/54 | 24/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Danicopan (TP1) (N=57) | Placebo (TP1) (N=29) | Danicopan-Danicopan (TP2) (N=55) | Placebo-Danicopan (TP2) (N=27) | Danicopan-Danicopan (LTE) (N=54) | Placebo-Danicopan (LTE) (N=26)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemolysis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Haemorrhagic diathesis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dieulafoy's vascular malformation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Stent-graft endoleak (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neutropenic sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Staphylococcal sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Body temperature increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Haemoglobin decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Paroxysmal nocturnal haemoglobinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Danicopan (TP1) (N=57) | Placebo (TP1) (N=29) | Danicopan-Danicopan (TP2) (N=55) | Placebo-Danicopan (TP2) (N=27) | Danicopan-Danicopan (LTE) (N=54) | Placebo-Danicopan (LTE) (N=26)
Haemolysis (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (4)
Neutropenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 3 (3) | 3 (3) | 0 (0) | 2 (2) | 1 (3)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 3 (12)
Nausea (Gastrointestinal disorders) | 5 (7) | 3 (3) | 1 (1) | 3 (3) | 3 (3) | 1 (3)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 3 (4) | 6 (7) | 2 (3) | 1 (2) | 2 (5)
Vomiting (Gastrointestinal disorders) | 3 (4) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (2)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Constipation (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 4 (4)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 2 (2)
Pyrexia (General disorders) | 3 (6) | 0 (0) | 7 (8) | 0 (0) | 13 (14) | 3 (5)
Chest discomfort (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Fatigue (General disorders) | 2 (2) | 1 (1) | 3 (3) | 1 (1) | 4 (6) | 1 (1)
Asthenia (General disorders) | 0 (0) | 4 (5) | 2 (2) | 2 (3) | 4 (4) | 4 (9)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 11 (11) | 7 (7)
Urinary tract infection (Infections and infestations) | 3 (3) | 1 (2) | 1 (1) | 1 (1) | 4 (4) | 2 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (4) | 2 (2) | 1 (1) | 1 (1) | 1 (3) | 1 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 4 (5) | 0 (0)
Headache (Nervous system disorders) | 6 (8) | 2 (2) | 6 (6) | 1 (1) | 8 (8) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 2 (2) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 3 (3)
Chromaturia (Renal and urinary disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (2) | 2 (2)
Hypertension (Vascular disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ear infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 1 (1)
Breakthrough haemolysis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 4 (5) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 7 (7) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 2 (2)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Contusion (Injury, poisoning and procedural complications) | 2 (2) | 3 (3) | 1 (3) | 1 (1) | 2 (2) | 0 (0)
Alanine aminotransferase increased (Investigations) | 3 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 3 (4) | 1 (1) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2022-08-08): https://cdn.clinicaltrials.gov/large-docs/65/NCT04469465/Prot_000.pdf
  • Statistical Analysis Plan (2022-08-10): https://cdn.clinicaltrials.gov/large-docs/65/NCT04469465/SAP_001.pdf